CLINICAL TRIAL: NCT05510778
Title: Effects of CharcoCaps® (Activated Charcoal) vs. Placebo on Intestinal Gas Production Assessed Using Breath Hydrogen and a Gastrointestinal Questionnaire
Brief Title: Effects of CharcoCaps® (Activated Charcoal) vs. Placebo on Intestinal Gas Production
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: DSE Healthcare Solutions (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of the College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRO-FY2022-9
Record Dates: First submitted 2021-12-08; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Intestinal Gas
Keywords: Charcocaps; Intestinal gas; Breath Hydrogen
MeSH Terms: conditions — Anthrax | interventions — Charcoal

STUDY DESIGN:
Intervention Model Description: double-blind, placebo controlled, cross-over
Who Masked: Participant, Investigator
Masking Description: Charcocaps and placebo capsules are similar in appearance and provided to investigators pre-masked (A and B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Charcocaps (Experimental): 2 capsules 15 minutes before meal and 2 additional capsules 2 hours after meal
  Interventions: Dietary Supplement: Charcocaps
- Placebo (Placebo Comparator): 2 capsules 15 minutes before meal and 2 additional capsules 2 hours after meal
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Charcocaps — 250 mg capsules containing Activated charcoal, Gelatin, Titanium Dioxide, and Carmine
  Arms: Charcocaps
Other: Placebo — capsules containing ~250 mg cellulose
  Arms: Placebo

SUMMARY:
Consumption of a high-fiber diet, often consisting of beans and vegetables, is recommended for improvements in overall health. Unfortunately, intake of the above-mentioned foods is often associated with a significant increase in intestinal gas production. In addition to gas, abdominal bloating, cramping, and associated symptoms can prove unacceptable-leading people to limit or abandon the consumption of bean-rich meals.

In an attempt to reduce gas formation and the ensuing symptoms, various anti-gas products have been developed and are sold on the market. One such non-prescription product is Beano, a solution of the enzyme alpha-galactosidase. In addition to alpha-galactosidase, activated charcoal has also been used successfully in some, but not all, studies and may be a good option for certain individuals.

CharcoCaps® is a branded form of activated charcoal that has been sold for several years.That said, no controlled studies have been conducted using CharcoCaps®. This study will investigate the effects of ingesting CharcoCaps® before and following the meal on the amount of gas produced, the number of flatus events, and associated symptoms of GI distress during the 6-hour post meal ingestion period.

DETAILED DESCRIPTION:
Consumption of a high-fiber diet, often consisting of beans and vegetables, is recommended for improvements in overall health. Adhering to such a dietary regimen is associated with weight management, as well as improvements in the blood lipid profile and glucose regulation (i.e., the prevention of type 2 diabetes). The end result is a lowering of the overall risk of cardio-metabolic disease .

Unfortunately, intake of the above mentioned foods is often associated with a significant increase in intestinal gas production, which has been suggested to be upwards of 10x that of a non-gas producing diet. This can be both uncomfortable and embarrassing when in social situations. In particular, flatus events are increased as a result of consumption of a bean-rich diet, with large volumes of flatus produced shortly after the ingestion of meals (within a few hours). In addition to flatus, abdominal bloating, cramping, and associated symptoms can prove unacceptable-leading people to limit or abandon the consumption of bean-rich meals.

In an attempt to reduce gas formation and the ensuing symptoms, various anti-gas products have been developed and are sold on the market. One such non-prescription product is Beano, a solution of the enzyme alpha-galactosidase. This product has been reported to effectively lower gas production (as evidenced by flatus events) following the consumption of a meatless chili meal, with the greatest improvements noted between 4-6 hours post meal ingestion.

In addition to alpha-galactosidase, activated charcoal has also been used successfully in some, but not all, studies and may be a good option for certain individuals. Activated charcoal is a fine, odorless powder formed from the destructive distillation of various organic materials, treated with substances such as steam or other chemicals at very high temperatures to increase its absorptive power. This agent is often described as a "rigid sponge" and has the ability to absorb many chemical substances, including gases. In fact, some have suggested that adding charcoal inside the seat cushions on airplanes may improve the flight experience for passengers, as released gas could be captured by the charcoal within the seats and reduce the odor.

CharcoCaps® is a branded form of activated charcoal that has been sold for several years, is widely available (e.g., Amazon, Walgreens, CVS), and has received excellent reviews from end users with regards to its ability to reduce intestinal gas production. That said, no controlled studies have been conducted using CharcoCaps®. Therefore, the following study will be conducted using a double-blind, placebo controlled, cross-over design to determine the impact of CharcoCaps® to reduce gas production and associated symptoms following the ingestion of a bean-rich meal. The investigators hypothesize that ingestion of CharcoCaps® before and following the meal will reduce the amount of gas produced, the number of flatus events, as well as associated symptoms of GI distress during the 6-hour post meal ingestion period.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of at least one of the following symptoms after eating meals rich in complex carbohydrates (such as beans):

  1. Abdominal bloating/pain/cramps
  2. Flatulence/gas
* Willing to consume a meatless chili meal and steamed broccoli
* No consumption of alcohol-containing beverages within 24 hours of testing
* No consumption of caffeine-containing beverages within 24 hours of testing
* No strenuous exercise within 24 hours of testing
* Be able to fast overnight (>10 hrs)

Exclusion Criteria:

* Diagnosed GI condition
* Diabetic
* Pregnant/lactating
* Self-reported active infection or illness of any kind
* Tobacco product user
* Hypersensitivity or allergy to any component of the supplement or chili (Activated charcoal, Gelatin, Titanium Dioxide, and Carmine, black beans, kidney beans, pinto beans, tomato puree, bell peppers, onion, sweet potato, chili powder, onion powder, garlic powder, salt, pepper, cumin, oregano, broccoli)
* Taking any anti-gas, or anti-flatulence medication or dietary supplements, or if taking only non-prescribed supplements/mediations, not willing to cease use of them during study period
* A regular consumer of bean meals (no more than once weekly)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Breath Hydrogen | 0 minutes before chili meal consumed (baseline)
  Hydrogen measured in exhale using H2 Check Analyzer
Breath Hydrogen | 30 minutes post meal consumption
  Hydrogen measured in exhale using H2 Check Analyzer
Breath Hydrogen | 60 minutes post meal consumption
  Hydrogen measured in exhale using H2 Check Analyzer
Breath Hydrogen | 90 minutes post meal consumption
  Hydrogen measured in exhale using H2 Check Analyzer
Breath Hydrogen | 120 minutes post meal consumption
  Hydrogen measured in exhale using H2 Check Analyzer
Breath Hydrogen | 150 minutes post meal consumption
  Hydrogen measured in exhale using H2 Check Analyzer
Breath Hydrogen | 180 minutes post meal consumption
  Hydrogen measured in exhale using H2 Check Analyzer
Breath Hydrogen | 210 minutes post meal consumption
  Hydrogen measured in exhale using H2 Check Analyzer
Breath Hydrogen | 240 minutes post meal consumption
  Hydrogen measured in exhale using H2 Check Analyzer
Breath Hydrogen | 270 minutes post meal consumption
  Hydrogen measured in exhale using H2 Check Analyzer
Breath Hydrogen | 300 minutes post meal consumption
  Hydrogen measured in exhale using H2 Check Analyzer
Breath Hydrogen | 330 minutes post meal consumption
  Hydrogen measured in exhale using H2 Check Analyzer
Breath Hydrogen | 360 minutes post meal consumption
  Hydrogen measured in exhale using H2 Check Analyzer
Gastrointestinal Symptoms Questionnaire | baseline
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Gastrointestinal Symptoms Questionnaire | 30 minutes post meal consumption
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Gastrointestinal Symptoms Questionnaire | 60 minutes post meal consumption
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Gastrointestinal Symptoms Questionnaire | 90 minutes post meal consumption
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Gastrointestinal Symptoms Questionnaire | 120 minutes post meal consumption
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Gastrointestinal Symptoms Questionnaire | 150 minutes post meal consumption
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Gastrointestinal Symptoms Questionnaire | 180 minutes post meal consumption
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Gastrointestinal Symptoms Questionnaire | 210 minutes post meal consumption
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Gastrointestinal Symptoms Questionnaire | 240 minutes post meal consumption
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Gastrointestinal Symptoms Questionnaire | 270 minutes post meal consumption
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Gastrointestinal Symptoms Questionnaire | 300 minutes post meal consumption
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Gastrointestinal Symptoms Questionnaire | 330 minutes post meal consumption
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Gastrointestinal Symptoms Questionnaire | 360 minutes post meal consumption
  Questionnaire that subject self-report the severity of gastrointestinal symptoms using a scale of 0 (no symptoms) to 10 (severe symptoms) for Bloating, Flatulence, Abdominal Rumblings, Abdominal Pain/Cramping, Stomach Fullness, Nausea, and Overall physical discomfort
Flatus events | baseline
  Self-reported number of flatus events each hour
Flatus events | 60 minutes post meal consumption
  Self-reported number of flatus events each hour
Flatus events | 120 minutes post meal consumption
  Self-reported number of flatus events each hour
Flatus events | 180 minutes post meal consumption
  Self-reported number of flatus events each hour
Flatus events | 240 minutes post meal consumption
  Self-reported number of flatus events each hour
Flatus events | 300 minutes post meal consumption
  Self-reported number of flatus events each hour
Flatus events | 360 minutes post meal consumption
  Self-reported number of flatus events each hour

SECONDARY OUTCOMES:
Concluding Questionnaire | 60 minutes post meal consumption
  Questionnaire where subjects provide written feedback on their perceptions of the assigned condition

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No